CLINICAL TRIAL: NCT04659135
Title: ASCO Survey on Coronavirus Disease 2019 (COVID-19) in Oncology (ASCO) Registry
Brief Title: ASCO Survey on COVID-19 in Oncology (ASCO) Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00014181
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms; Coronavirus
Keywords: Cancer
MeSH Terms: conditions — Neoplasms; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The American Society of Clinical Oncology (ASCO) Survey on Coronavirus 2019 (COVID-19) in Oncology Registry (ASCO Registry) aims to help the cancer community learn more about the patterns of symptoms and severity of COVID-19 among patients with cancer, as well as how COVID-19 is impacting the delivery of cancer care and patient outcomes. The ASCO Registry collects both baseline and follow-up data on how the virus impacts cancer care and cancer patient outcomes during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Rationale:

The COVID-19 Pandemic presents a unique opportunity to capture information on how a disease outbreak affects delivery of high-quality cancer care. ASCO is providing the means for the oncology community to rapidly submit data that will inform both current cancer care and provide information to help guide decision-making for future disease outbreaks. While other entities have launched COVID-19 cancer registries, ASCO's registry collects information about patients undergoing treatment for cancer and with confirmed COVID-19 infection based on a positive test. Unlike other registries, ASCO's registry collects follow-up information on both COVID-19 disease and cancer outcomes at 30-day intervals for the first 90 days and 90-day intervals thereafter up to one year after COVID-19 diagnosis.

Project Objectives:

Capture and describe cancer and COVID-19 status at COVID-19 diagnosis, and cancer and COVID-19 outcomes of patients with cancer and COVID-19 from participating cancer practices/institutions. Data collected includes treatment approaches, cancer status, changes to cancer treatment plans in patients with confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, status of COVID-19 infection (e.g., severity of symptoms, need for ventilator, hospitalization, etc.) and cancer (e.g., cancer progression, treatment-related changes/modifications, etc.).

Research Objectives:

Objective 1: Describe the distribution of symptoms and severity of COVID-19 among patients with cancer (on active treatment or on adjuvant treatment within 12 months after surgical resection) who have confirmed infection of SARS-CoV-2 •Objective 1.1: Describe distribution of symptoms and severity of COVID-19 stratified according to demographic characteristics, including age, cancer type, cancer extent, race, ethnicity, geography, type of therapy received, smoking status, comorbidities, etc.

•Objective 1.2: Identify characteristics independently associated with severity of COVID-19 in cancer patients.

Objective 2: Examine SARS-CoV-2 viral infection outcomes (ongoing, recovery, hospitalized, not in ICU; hospitalized in ICU; placed on ventilator; death due to COVID-19 disease complications) and cancer outcomes (stable, response to treatment, progression, delayed treatment, treatment discontinued, and death)

* Objective 2.1: Stratify patients with SARS-CoV-2 viral infection according to characteristics described in Objective 1.1 to examine whether any of the characteristics are independently associated with COVID-19 and/or cancer outcomes
* Objective 2.2: Examine the relationship between SARS-CoV-2 viral infection outcomes and cancer outcomes and whether SARS-CoV-2 viral infection outcomes are independently associated with cancer outcomes

Objective 3: To describe effects of the COVID-19 pandemic on cancer practices in the U.S., including changes in staffing and resource availability, priorities for patient care, and modification of interactions between care providers and patients (including use of telemedicine)

Eligibility Criteria:

The registry collects data about patients with a cancer diagnosis who have a confirmed SARS-CoV-2 infection and are being treated at participating cancer practices/institutions within the United States. Patients in one of the four categories are eligible:

1. Patients with a new cancer diagnosis and in the process of cancer staging and/or receipt of initial cancer therapy
2. Patients with clinically evident cancer receiving anti-cancer treatment,
3. Patients who are disease free, but receiving any type of adjuvant therapy within 1 year following surgical resection (including hormonal treatments), and
4. Patients with clinically evident cancer receiving supportive care only.

Statistical Considerations and Reporting:

ASCO's Center for Research and Analytics (CENTRA) reports via a data dashboard (https://www.asco.org/covid-resources/asco-registry/data-dashboard) to the general cancer community key characteristics of patients in the Registry. ASCO also submits abstracts for presentation and manuscripts for publication. Reports summarize overall data and stratified by patient characteristics, such as disease sites and stage, age and comorbidities. Reports or publications will also include cancer treatment delay and discontinuation of cancer treatments including surgery, radiation and drug-based therapies, due to the patient's COVID-19 disease and to other factors, with stratification by other variables as described above. Changes in practice patterns of care, staffing, resources, and interactions with patients will also be evaluated and summarized.

As there is no hypothesis testing planned, there is no required sample size and providing reports also provided to other registries, with cumulative information, will not affect validity of results. Confidence intervals will be provided where appropriate to demonstrate precision of estimates.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive diagnosis
* One of the following;

  1. Patient has active cancer at the time of COVID-19 diagnosis OR
  2. Patient has been cancer-free for less than 12 months AND receiving adjuvant therapy at the time of COVID-19 diagnosis

Exclusion Criteria:

* COVID-19 suspected, but no positive test result
* Patient is a cancer-free not receiving any anti-cancer or adjuvant treatment
* Patient is receiving adjuvant therapy, but has been cancer-free for up to 12 months at the time of COVID-19 diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a cancer diagnosis who have a confirmed SARS-CoV-2 infection and are being treated for their cancer at participating cancer practices/institutions within the United States
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2020-04-19 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Changes to Cancer Treatments | 24 months
  Treatments: Yes vs. no response to changes in reported treatment administration for anti-cancer therapeutics

SECONDARY OUTCOMES:
All-cause mortality at 30 days | 30 days
  Any patient deaths that occurred as measured by number of days after COVID-19 diagnosis
COVID-19 Symptoms | 24 months
  Yes vs. no response to reported COVID-19 symptoms
COVID-19 Treatments | 24 months
  Yes vs. no response to reported treatment administration for anti-COVID-19 therapeutics
Patient vital status | 24 months
  Alive vs. dead up to 24 months from COVID-19 diagnosis
Overall survival | 24 months
  Time to event endpoint measured as the time from covid-19 dx to death, censored at the last time patient was known to be alive if there is no death date provided.
Patient cancer status (for patients who had active cancer at covid-19 dx) | 24 months
  Categorical variable of cancer status, compared to time at COVID-19 diagnosis (stable, responding to therapy, progressed). This will be measured over time (longitudinally) and can take different values for the same patient at different time points.
Patient cancer status (for patients who are disease-free at COVID-19 diagnosis) | 24 months
  An indicator (yes v no) of whether the patients cancer has relapsed since COVID-19 diagnosis. This will be measured over time (longitudinally) and can take different values for the same patient at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Gralow, MD, Principal Investigator — American Society of Clinical Oncology; Suanna S Bruinooge, MPH, Study Director — American Society of Clinical Oncology; Elizabeth Garrett-Mayer, PhD, Study Director — American Society of Clinical Oncology
Locations (77):
- United States (77):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - Anchorage Oncology Center, Anchorage, Alaska
  - AIS Cancer Center, Bakersfield, California
  - Long Beach Memorial Medical Center, Fountain Valley, California
  - Orange Coast Medical Center, Fountain Valley, California
  - Saddleback Memorial Medical Center, Fountain Valley, California
  - Helen Diller Family Comprehensive Cancer Center, UCSF, San Francisco, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - PIH Health, Whittier, California
  - Hartford HealthCare Cancer Institute, Hartford, Connecticut
  - Day Kimball Healthcare, Putnam, Connecticut
  - Bayhealth Medical Center, Dover, Delaware
  - Florida Precision Oncology, A Division of 21st Centry Oncology, Fort Myers, Florida
  - Florida Cancer Specialists - Sarah Cannon Research Institute, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Cancer Center of Middle Georgia, LLC, Dublin, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - OSF Little Company of Mary Hospital, Evergreen Park, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Edward-Elmhurst Healthcare, Naperville, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Quincy Medical Group Cancer Institute, Quincy, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Michiana Hematology Oncology, Mishawaka, Indiana
  - Midwest Oncology Associates - Sarah Cannon Research Institute, Overland Park, Kansas
  - University of Kansas Medical Center, Westwood, Kansas
  - Baptist Health Madisonville, Madisonville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital Cancer Institute, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Great Lakes Cancer Management Specialists, Grosse Pointe Woods, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Boone Hospital Center, Columbia, Missouri
  - Mosaic Cancer Care, Saint Joseph, Missouri
  - Nebraska Hematology Oncology, Lincoln, Nebraska
  - Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Bayonne Medical Center, Bayonne, New Jersey
  - CarePoint Health - Christ Hospital, Jersey City, New Jersey
  - Penn Medicine, Princeton Health, Plainsboro, New Jersey
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute Atrium Health, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Carteret Health Care, Morehead City, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - TriCounty Hematology and Oncology, Massillon, Ohio
  - Columbia Memorial Hospital, Astoria, Oregon
  - Samaritan Health Services Corvallis, Corvallis, Oregon
  - Penn Medicine, Lancaster General Health, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lexington Oncology, West Columbia, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Kirkland Cancer Center, Jackson, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The START Center for Cancer Care, San Antonio, Texas
  - University of Texas, Health Science Center, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Augusta Health, Fishersville, Virginia
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - PeaceHealth, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
ASCO is making deidentified Registry data available to researchers (both those at Registry sites and those not involved with the Registry) who submit a qualified research proposal for further analysis. ASCO reviews requests for Registry data from individuals and entities that submit a research proposal that complies with ASCO's requirements for data access. ASCO will promote access to information for projects that address the needs of patients with cancer, including marginalized populations and communities. ASCO will promote authenticity, quality, reliability and integrity of information and analyses. ASCO will promote fair access and efficiency in the use and sharing of ASCO Information within the bounds of this Policy.
Supporting Information: Study Protocol, SAP
Time Frame: First Quarter 2022
Access Criteria: Completion of a satisfactory Research Project Proposal Application, as discussed on the ASCO Data Library website
URL: https://old-prod.asco.org/research-data/asco-data-library

REFERENCES:
- [Background] Mullangi S, Aviki EM, Hershman DL. Reexamining Social Determinants of Health Data Collection in the COVID-19 Era. JAMA Oncol. 2022 Dec 1;8(12):1736-1738. doi: 10.1001/jamaoncol.2022.4543. PMID 36301554
- [Result] Kurbegov D, Bruinooge SS, Lei XJ, Kirkwood MK, Dickson N, Hattiangadi T, Mileham KF, Patrick A, Williams JH, Kaltenbaugh M, Gralow JR, Garrett-Mayer E. Rate of COVID-19 vaccination among patients with cancer who tested positive for severe acute respiratory syndrome-coronavirus 2: Analysis of the American Society of Clinical Oncology Registry. Cancer. 2023 Jun 1;129(11):1752-1762. doi: 10.1002/cncr.34726. Epub 2023 Mar 15. PMID 36920457
- [Result] Mileham KF, Bruinooge SS, Aggarwal C, Patrick AL, Davis C, Mesenhowski DJ, Spira A, Clayton EJ, Waterhouse D, Moore S, Jazieh AR, Chen RC, Kaltenbaugh M, Williams JH, Gralow JR, Schilsky RL, Garrett-Mayer E. Changes Over Time in COVID-19 Severity and Mortality in Patients Undergoing Cancer Treatment in the United States: Initial Report From the ASCO Registry. JCO Oncol Pract. 2022 Apr;18(4):e426-e441. doi: 10.1200/OP.21.00394. Epub 2021 Oct 25. PMID 34694907
- [Result] Llanos AAM, Ashrafi A, Ghosh N, Tsui J, Lin Y, Fong AJ, Ganesan S, Heckman CJ. Evaluation of Inequities in Cancer Treatment Delay or Discontinuation Following SARS-CoV-2 Infection. JAMA Netw Open. 2023 Jan 3;6(1):e2251165. doi: 10.1001/jamanetworkopen.2022.51165. PMID 36637818
- [Result] Mullangi S, Aviki EM, Chen Y, Robson M, Hershman DL. Factors Associated With Cancer Treatment Delay Among Patients Diagnosed With COVID-19. JAMA Netw Open. 2022 Jul 1;5(7):e2224296. doi: 10.1001/jamanetworkopen.2022.24296. PMID 35900758

DOCUMENTS (1):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04659135/Prot_000.pdf